CLINICAL TRIAL: NCT01015001
Title: A Pilot Double-blind Sham-controlled Trial of Repetitive Transcranial Magnetic Stimulation for Patients With Refractory Schizophrenia Treated With Clozapine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: FIPE, Hospital de Clínicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06382
Record Dates: First submitted 2009-11-10; First posted 2009-11-17 (Estimated); Last update posted 2010-08-12 (Estimated); Status verified 2010-08

CONDITIONS: Schizophrenia; Auditory Hallucinations
Keywords: refractory schizophrenia; rTMS; auditory hallucinations
MeSH Terms: conditions — Schizophrenia; Hallucinations; Schizophrenia, Treatment-Resistant | interventions — Transcranial Magnetic Stimulation; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active rTMS (Active Comparator): 1Hz rTMS sessions applied to the left temporoparietal cortex of the subjects
  Interventions: Procedure: Active rTMS x sham (placebo) rTMS; Procedure: (1Hz) rTMS applied over the left temporoparietal cortex
- Sham rtms (Placebo Comparator): Same number of pulses but applied with and angled coil (90 degrees) and placed over the fronto´temporal region
  Interventions: Procedure: Active rTMS x sham (placebo) rTMS; Procedure: sham rTMS

INTERVENTIONS:
Procedure: Active rTMS x sham (placebo) rTMS — Seventeen right-handed patients with DSM-IV TR diagnosis of schizophrenia were randomized in two groups. One arm received 20 sessions of 20 minutes each of low-frequency (1Hz) rTMS applied over the left temporoparietal cortex (LTPC).
  The other arm received sham (placebo) stimulation over the LTPC for the same period of time. All patients were considered as having refractory schizophrenia and in use of at least 400mg/day of clozapine and referred auditory hallucinations.
  Other Names: EMTr
Procedure: sham rTMS — same coil, same number of pulses but using an angled coil(90degres) over the frontotemporal region
  Other Names: Sham
  Arms: Sham rtms
Procedure: (1Hz) rTMS applied over the left temporoparietal cortex — 20 sessions lasting 20 minutes each of low-frequency (1Hz) rTMS applied over the left temporoparietal cortex (LTPC).
  Arms: Active rTMS

SUMMARY:
The primary outcome of this study is to evaluate the effects of low frequency subthreshold repetitive Transcranial Magnetic Stimulation applied to the left temporoparietal cortex of patients with refractory schizophrenia on the severity of auditory hallucinations.

The secondary outcome is to evaluate the effects of the same rTMS protocol on quality of life, functionality and general psychopathology.

DETAILED DESCRIPTION:
Seventeen patients with DSM-IV TR diagnosis of schizophrenia were randomized in two groups. First group received 20 sessions of 20 minutes each of low-frequency (1Hz) rTMS applied over the left temporoparietal cortex (LTPC).

Second group received sham (placebo) stimulation over the LTPC for the same period of time. All patients were considered as having refractory schizophrenia and in use of at least 400mg/day of clozapine and refering auditory hallucinations occuring at least 5 times a day.

ELIGIBILITY:
Inclusion Criteria:

* Patients with DSM IV TR diagnose of schizophrenia with treatment-resistant auditory hallucinations.
* Use of at least 400mg/day of clozapine
* Men and women from 18 to 65 years old
* Fertile women must be using adequate contraceptive method
* BPRS score of at least 27

Exclusion Criteria:

* Suicide risk
* Patients with epilepsy, brain surgery and/or head trauma in the past, use of cardiac pace maker or metalic clip in the head
* Diagnose of substance abuse/dependance
* Severe uncontrolled organic disease that may interfere in the patient´s participation in the study
* Any other reason that, in the investigator´s opinion, might interfere with the patient´s participation in the study, such as non compliance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the effects of low frequency repetitive Transcranial Magnetic Stimulation applied over the left temporoparietal cortex of refractory schizophrenic patients on the severity of auditory hallucinations. | 2 years

SECONDARY OUTCOMES:
The secondary outcomes are to evaluate the effects of the same rTMS protocol on their quality of life, functionality and general psychopathology. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Danilo Jesus, Psychiatrist, Principal Investigator — Hospital de Clinicas de Porto Alegre; Paulo B Abreu, phd, Study Director — HCPorto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil